CLINICAL TRIAL: NCT03051165
Title: Effect of Upper Airway Stimulation on Vascular Function in Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to funding issues.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Raj Dedhia, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00088693
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Cardiovascular Disease; Pulmonary Medicine; Hypoglossal Nerve Stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: All participants will undergo the intervention of temporary treatment withdrawal to examine cardiac measurements before treatment, during treatment, and after cessation.
Masking Description: Interpretation of all tests (sleep tests, ambulatory blood pressure monitoring, vascular test and blood tests) will be done by an outcomes assessor who is blinded to whether treatment is active or withheld at the time of testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypoglossal Nerve Stimulation Treatment Withdrawal (Other): Recipients of hypoglossal nerve stimulation (HGNS) who agree to participate in the study will have additional tests done to monitor cardiovascular responses to HGNS therapy and the temporary withdrawal of treatment.
  Interventions: Device: Hypoglossal Nerve Stimulation Treatment Withdrawal

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation Treatment Withdrawal — After 90 days of hypoglossal nerve stimulation (HGNS), therapy will be discontinued for 30 days before being reactivated.
  Other Names: HGNS

SUMMARY:
This study will evaluate the effect of hypoglossal nerve stimulation (HGNS) on different measures of cardiovascular function in patients with obstructive sleep apnea (OSA). People with OSA who have undergone implantation of the hypoglossal nerve stimulator at the study site will be told about the study at their 2-week post-operative appointment. Those who decide to participate will have blood drawn and vascular function measurements taken before HGNS activation, during treatment, and after a temporary treatment withdrawal period. Following the 30-day period of treatment withdrawal, the HGNS therapy will be reactivated.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), the repetitive collapse of the upper airway during sleep, represents a growing individual and public health concern. This disease negatively impacts patients' sleep quality and daytime function, including an increased risk of motor vehicle accidents. Several large, longitudinal cohorts have consistently demonstrated deleterious effects of OSA on cardiovascular health, including elevated rates of incident hypertension, myocardial infarction and cerebrovascular accidents. The link between OSA and cardiovascular consequences can be largely explained by autonomic imbalance during repeated episodes of nocturnal airway obstruction. Compared to those without OSA, people with OSA have increased sympathetic activity when awake, with further elevation of both sympathetic activity and blood pressure during sleep. Multiple physiologic mechanisms are responsible for these autonomic changes during obstructive episodes including the interaction of baroreceptors, chemoreceptors and respiratory afferent receptors.

Positive airway pressure (PAP) serves as a pneumatic stent for the airway, maintaining airway patency and normoxia. PAP therapy has demonstrated consistent, meaningful reductions in sympathetic overactivity during wake and sleep. Although PAP therapy is highly efficacious, fewer than 50% of patients are adequately treated due to adherence difficulty. In 2014, the Federal Drug Administration approved hypoglossal nerve stimulation (HGNS) for the treatment of patients with moderate-severe OSA who are unable to adequately use PAP. This therapy has demonstrated stable, marked improvement in key polysomnography indices, sleepiness measures and functional outcomes, however, no study has examined cardiovascular endpoints of HGNS therapy in OSA patients.

The aim of this study is to evaluate the effect of HGNS therapy on autonomic and vascular function before, during and after treatment for OSA with HGNS. People who have undergone implantation of the hypoglossal nerve stimulator at the study site will be told about the study at their 2-week post-operative appointment. Those who decide to participate in the study will have blood drawn and vascular function measurements taken before the HGNS device is activated, during treatment, and after a temporary treatment withdrawal period. The researchers hypothesize that all aforementioned measurements will be significantly improved following HGNS therapy and return to baseline values following a therapy withdrawal period.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Able to give informed consent
* Have undergone implantation of hypoglossal nerve stimulator (HGNS) by the principal investigator of this study. HGNS inclusion criteria per FDA are as follows:

  * Apnea-hypopnea index (AHI) of 20 or more from recent sleep test
  * Unable to use positive airway pressure therapy
  * Body Mass Index (BMI) < 32 kg/m2
  * Without circumferential collapse on drug-induced sedated endoscopy

Exclusion Criteria:

* Active smokers
* Unstable and untreated coronary or peripheral artery disease
* Use of alpha-blockers
* Severe and inadequately controlled arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Dedhia, MD, Principal Investigator — Emory University
Locations (1):
- Emory Sleep Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Sleep Center in Atlanta, Georgia. Enrollment began on 11/21/2016 and the study was terminated early on 12/14/2017.
Groups:
- Hypoglossal Nerve Stimulation Treatment Withdrawal: Recipients of hypoglossal nerve stimulation (HGNS) who consented to have temporary withdrawal of treatment.
Period: Overall Study
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Started | 13
Completed Some Baseline Assessments (Baseline assessments refer to clinical assessments; demographic information was collected for all.) | 1
Completed Some Day 105 Assessments (Day 105 assessments occur just prior to HGNS treatment withdrawal.) | 1
Began HGNS Treatment Withdrawal | 0
Completed Some Day 137 Assessments (Day 137 assessments occur after 30 days of HGNS treatment withdrawal.) | 0
Completed | 0
Not Completed | 13
Not completed — Withdrawal by Subject | 1
Not completed — Early termination of study | 12

BASELINE CHARACTERISTICS:
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Peripheral Arterial Tonometry (PAT)
Description: Peripheral arterial tonometry (PAT) is a method for measuring endothelial dysfunction in a non-invasive way. Blood flow is measured in the fingertips following compression with an inflatable cuff on the upper arm. Participants will lay on their backs with a probe placed on the finger of each hand. The probes are attached to a computer that records finger blood flow. The finger probes will continuously record the blood flow in the fingertips for 10 minutes
Time Frame: Baseline, Day 105, Day 137
Population: PAT assessment was not performed for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Flow Mediated Dilation
Description: Flow mediated dilation is a method to assess endothelial function using an ultrasound device to take measurements of the artery at the elbow. Blood vessel diameter is measured before and after blood pressure cuff release and flow mediated dilation is the percent of change between the baseline and post cuff release measurements. A lower measurement of dilation corresponds with an increased risk for cardiovascular events.
Time Frame: Baseline, Day 105, Day 137
Population: One participant completed the flow mediated dilation assessment at Baseline and Day 105.
Measure: Mean (Standard Deviation); unit: percentage of baseline arterial diameter
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 1
percentage of baseline arterial diameter
  Baseline (before initial device activation) | 2.23 (0.0)
  Day 105 (after 90 days of device activation) | 4.75 (0.0)

3. Secondary Outcome: Change in Peripheral Arterial Stiffness
Description: Recordings of blood flow through the artery in the wrist will be obtained with application of a probe applied to the skin. Participants will be seated or lying down for this test which takes approximately 10 minutes. Increased arterial stiffness is associated with an increased risk of cardiovascular events.
Time Frame: Baseline, Day 105, Day 137
Population: Peripheral arterial stiffness assessment was not performed for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in 24-hour Ambulatory Blood Pressure
Description: To measure 24-hour ambulatory blood pressure, participants wear a watch like device on one arm which records blood pressure throughout the day.
Time Frame: Baseline, Day 105, Day 137
Population: One participant completed the 24-hour ambulatory blood pressure Baseline assessment.
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 1
mm/Hg
  Baseline Visit Systolic Blood Pressure | 133 (0.0)
  Baseline Visit Diastolic Blood Pressure | 67 (0.0)

5. Secondary Outcome: Change in C-reactive Protein
Description: To assess changes in the serum biomarker profile, blood will be collected from participants to be stored for future analyses of a variety of biochemical factors related to cardiovascular function. C-reactive protein is produced by the liver and increased concentrations are found when inflammation is present in the body.
Time Frame: Baseline, Day 105, Day 137
Population: Blood for serum biomarker assessments was not collected for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Fibrin Degradation Products
Description: To assess changes in the serum biomarker profile, blood will be collected from participants to be stored for future analyses of a variety of biochemical factors related to cardiovascular function. Fibrin degradation products are produced by of clot degeneration. Plasma fibrin degradation products increase following clot formation.
Time Frame: Baseline, Day 105, Day 137
Population: Blood for serum biomarker assessments was not collected for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Heat Shock Protein 70 (HSP70)
Description: To assess changes in the serum biomarker profile, blood will be collected from participants to be stored for future analyses of a variety of biochemical factors related to cardiovascular function. Heat shock protein 70 (HSP70) is a stress protein. Heat shock proteins increase in response to stress conditions such as inflammation and infection.
Time Frame: Baseline, Day 105, Day 137
Population: Blood for serum biomarker assessments was not collected for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in High Sensitivity Cardiac Troponin (HS-troponin)
Description: To assess changes in the serum biomarker profile, blood will be collected from participants to be stored for future analyses of a variety of biochemical factors related to cardiovascular function. Elevated high sensitivity cardiac troponin (HS-troponin) indicates injury to the heart.
Time Frame: Baseline, Day 105, Day 137
Population: Blood for serum biomarker assessments was not collected for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Soluble Urokinase-type Plasminogen Activator Receptor (suPAR)
Description: To assess changes in the serum biomarker profile, blood will be collected from participants to be stored for future analyses of a variety of biochemical factors related to cardiovascular function. Soluble urokinase-type plasminogen activator receptor (suPAR) is a marker for disease status by indicating the degree of activation of the immune system. Higher concentrations indicate inflammation and are associated with an increased risk of mortality.
Time Frame: Baseline, Day 105, Day 137
Population: Blood for serum biomarker assessments was not collected for any participants at any study visit.
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on study participants from the time of consent through reactivation of HGNS therapy (Day 1 through Day 137).
Arm/Group | Hypoglossal Nerve Stimulation Treatment Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03051165/Prot_SAP_000.pdf